CLINICAL TRIAL: NCT04326192
Title: Brown Adipose Tissue Activation by Spinal Cord Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kim J. Burchiel, Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020197
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Pain, Back; Obesity, Morbid; Type 2 Diabetes
Keywords: Obesity; Diabetes
MeSH Terms: conditions — Back Pain; Obesity, Morbid; Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All subjects (Experimental): All subjects will have two PET/CT scans on days 3 and 5 after SCS electrode implantation: (1) Baseline and (2) SCS-activated. Other than SCS activation, both studies will be conducted under identical conditions. For the first scan, subjects will be randomly assigned to either a baseline (no SCS during PET/CT) or with SCS during PET/CT prior to the day of their first scan. The second scan will complete the sequence with either a baseline or SCS-activated scan, as randomized.
  Interventions: Device: Research electrode

INTERVENTIONS:
Device: Research electrode — A second electrode will be placed percutaneously by Tuohy needle in the epidural space at the same time as the SCS trial implant; at lateral T1-2 area randomly assigned to the left or right side of the lateral epidural space, at the time of the procedure. Placement of electrodes is not experimental, but the placement of a second electrode is a research-driven procedure.

SUMMARY:
The objective of this study is to investigate and utilize spinal cord stimulation (SCS) as an effective approach to eliciting weight loss and potentially alleviating Type 2 diabetes mellitus (DM), as evidenced by increasing metabolism of adipose tissue.

DETAILED DESCRIPTION:
This research study aims to investigate possible activation of brown adipose tissue (BAT) metabolism by upper thoracic spinal cord stimulation (SCS). We believe that our multidisciplinary research team presents a unique opportunity to test whether SCS can activate BAT metabolism, as tested during a routine screening procedure for spinal cord stimulation (SCS) for pain control. Our marker for BAT activation is 18F-fluorodeoxyglucose (FDG) - positron emission tomography (PET), which has previously been used to gauge cold-evoked BAT activation, and other studies of BAT in humans. We believe this proof-of-concept study could pave the way for a new therapeutic modality for the treatment of morbid obesity, and Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 21-70 years
2. Persistent neuropathic leg and back pain
3. Subjects who are already planning to undergo SCS for pain
4. Subjects who have not received a prior SCS trial for pain
5. Subjects with a BMI of 25-45, using formula; weight (lb) / [height (in)]2 x 703

Exclusion Criteria:

1. Not considering SCS for pain
2. Forensic patient
3. Taking beta blockers
4. Weight change > 5% within last 3 months
5. Habitual tobacco use
6. Habitual excessive alcohol use
7. Pregnancy
8. Decisionally impaired adults
9. Children
10. Neonates
11. Subjects with a BMI of <25 or >45

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 1 week
  Maximum standardized uptake value (SUVmax) of bilateral cervical and supraclavicular regions during SCS activation, in comparison to baseline imaging

SECONDARY OUTCOMES:
Ipsi- and contralateral BAT during SCS-activation | 1 week
  A comparison of ipsi- and contralateral BAT during SCS-activation. PET/CT images will be reconstructed as per standard clinical routine.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Burchiel, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No